# JSS Medical Research India Private Limited Data Management



## Statistical Analysis Plan

SOP Number: JSS-DM-BIS-01

Current Version Number: 1.0 Previous Version Number: None :None Document Date:06NOV2019

## STATISTICAL ANALYSIS PLAN

**Protocol Title:** A Multi-Center, Open-Label, Pharmacokinetic,

and Safety Study for Reduction in Fever or Management of Pain in Pediatric Subjects Aged

Birth to Six Months

**Protocol No.:** CPI-CL-022

**Protocol Date:** 01Jun2015

**SAP Version:** 1.0

**SAP Date:** 06NOV2019

#### **Prepared By:**

JSS Medical Research India Private Limited Data Management 6th Floor, Vatika Mindscapes (Tower B) Plot 12/2, Sector 27D Faridabad, Haryana India 121003

Telephone

Fax

#### **Sponsor:**

Sr. Vice President & Chief Development Officer Cumberland Pharmaceuticals Inc. 2525 West End Avenue, Suite 950 Nashville, TN 37203 USA

| Cumberland Pharmaceuticals Inc. | JSS Medical Resea | JSS PESPONSIVE PEUABLE RESULTS. | |
|---|---|---|---|
| Statistical Analysis Plan | | | |
| SOP Number:<br>JSS-DM-BIS-01 | Current Version<br>Number:1.0 | Previous Version Number:<br>None :None | ument<br>e:06NOV2019 |

#### **Sponsor Signature**

I hereby declare that I have reviewed the statistical analysis plan and agree to its form and content. In addition, I confirm that the outlined statistical analysis plan contains all relevant information for the data analysis to be performed in the Protocol No. CPI-CL-022 study by the Biostatistics Department.

| Date | | |
|-----------------------------|-----------------|------|
| Date Represented by: Date | | |
| Represented by: Date | Represented by: | |
| Represented by: Date | | Data |
| Date | | Date |
| Date | | |
| Date | | |
| | Represented by: | |
| Biostatistician | | Date |
| Biostatistician | | |
| Biostatistician | | |
| Biostatistician | | |
| | Biostatistician | |
| Date | | |

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

None: None

SOP Number: JSS-DM-BIS-01

Current Version Number: 1.0 Previous Version Number:

ber: Document
Date:06NOV2019

#### **Authorization Document**



| Cumberland |
|------------------------|
| <b>Pharmaceuticals</b> |
| Inc. |

# JSS Medical Research India Private Limited Data Management



## Statistical Analysis Plan

SOP Number:

JSS-DM-BIS-01

Current Version
Number:1.0

Previous Version Number:
None:None

Document
Date:06NOV2019

### **TABLE OF CONTENTS**

| LIST O | OF ABBREVIATIONS AND DEFINITION OF TERMS | 9 |
|--------|---------------------------------------------|----|
| 1.0 | INTRODUCTION | 10 |
| 2.0 | DESCRIPTION OF THE PROTOCOL | 10 |
| 2.1 | Protocol Number | 10 |
| 2.2 | Protocol Title | 10 |
| 2.3 | Date | 10 |
| 2.4 | Amendment | 10 |
| 3.0 | STUDY OBJECTIVES AND ENDPOINTS | 10 |
| 3.1 | Study Objectives | 10 |
| 3.1.1 | Primary Objectives | 10 |
| 3.1.2 | Secondary Objectives | 11 |
| 3.2 | End Points | 11 |
| 3.2.1 | Primary Pharmacokinetic Endpoints | 11 |
| 3.2.2 | Secondary (Safety) Endpoints | 11 |
| 4.0 | STUDY METHODS | 11 |
| 4.1 | Study Design and Plan | 11 |
| 4.2 | Study Initiation and Completion | 12 |
| 4.3 | Selection of Study Population | 12 |
| 4.3.1 | Screening Population (SCREEN) | 12 |
| 4.3.2 | Safety population | 12 |
| 4.3.3 | PK (Pharmacokinetics) -evaluable Population | 12 |
| 4.4 | Study Subject Group | 12 |
| 4.5 | Study Background | 12 |
| 4.6 | Study Rationale | 12 |

# JSS Medical Research India Private Limited Data Management



| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

| 4.7 | Schedule of Study Events | 13 |
|------|--------------------------------------------------------|----|
| 4.8 | Schedule of Visits and Procedures | 13 |
| 5.0 | GENERAL CONSIDERATIONS FOR STATISTICAL ANALYSIS | 14 |
| 5.1 | Sample Size Determination | 14 |
| 5.2 | Method of Treatment Assignment and Randomization | 14 |
| 5.3 | Methods for Withdrawals and Missing Data | 14 |
| 5.4 | Analysis Software | 15 |
| 6.0 | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | 15 |
| 6.1 | Demographics | 15 |
| 6.2 | Baseline and Screening Conditions | 15 |
| 6.3. | Baseline Medical History | 16 |
| 6.4 | Physical Examination | 16 |
| 7.0 | STATISTICAL ANALYSES | 16 |
| 7.1 | Primary Endpoint Analysis (Pharmacokinetic Parameters) | 16 |
| 7.2 | Secondary Endpoint Analysis | 16 |
| 8.0 | SAFETY AND TOLERABILITY ANALYSES | 17 |
| 8.1 | Adverse Events | 17 |
| 8.2 | Vital Signs | 17 |
| 8.3 | Concomitant Medication | 17 |
| 8.4 | Laboratory parameters | 17 |
| 9.0 | INTERIM ANALYSIS OR OTHER PLANNED ANALYSES | 18 |
| 10.0 | REPORTING CONVENTIONS | 18 |
| 10.1 | Reporting of Numeric Values | 18 |
| 11.0 | OUTPUT (TABLES, LISTINGS AND GRAPHS) CONSIDERATIONS | 18 |
| 12.0 | REFERENCES | 19 |
| APPE | ENDIX 1: SUMMARY OF STATISTICAL ANALYSIS | 20 |

# JSS Medical Research India Private Limited Data Management



| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

| 1.1 | TABLES | 20 |
|---|---|---|
| 14.1.1 | Subject Disposition | 20 |
| Table 14 | .1.1.1 Summary of Inclusion/Exclusion Criteria – All Screened (N=) | 20 |
| Table 14 | .1.1.2 Summary of Study Populations – All Enrolled (N=) | 21 |
| 14.1.2 | Demographics and Baseline Characteristics | 22 |
| Table 14 | .1.2.1 Summary of Subject Demographics-Safety Population (N=) | 22 |
| 14.1.3 | Medical History | 24 |
| Table 14 | .1.3.1 Summary of Medical History by SOC and PT-Safety Population (N=) | 24 |
| 14.1.4 | Physical Examination | 25 |
| Table 14 | .1.4.1 Summary of Physical ExaminationSafety Population (N=) | 25 |
| 14.2 | Efficacy Analysis | 26 |
| 14.2.1 | Primary Efficacy Analysis | 26 |
| Table 14 | .2.1.1 Summary of Statistics of Pharmacokinetics (PK) Parameters-PK Population(N=) | 26 |
| 14.2.2 | Secondary Analysis (Safety Endpoint) | 29 |
| Table 14 | .2.2.1 Summary of Overall Treatment Emergent Adverse Events -Safety Population (N=) | 29 |
| Table 14 | .2.2.2. Summary of Treatment Emergent Adverse Events by System Organ Class (SOC) and Preferred Term (PT)- Safety Population (N=) | 31 |
| Table 14 | .2.2.3 Summary of Vital Signs – Safety Population (N=) | 32 |
| Table 14 | .2.2.4 Summary of Coagulation Assessments – Safety Population (N=) | 34 |
| Table 14 | .2.2.5 Summary of Haematology – Safety Population (N=) | 36 |
| Table 14 | .2.2.6 Summary of Chemistry – Safety Population (N=) | 38 |
| 14.3 | Safety Analysis | 40 |
| 14.3.1 A | DVERSE EVENTS | 40 |
| Table 14 | .3.1.1 Summary of Overall Adverse Events -Safety Population (N=) | 40 |
| Table 14 | .3.1.2. Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) - Safety Population(N=) | 42 |

# JSS Medical Research India Private Limited Data Management



| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

| Table 14.3.1.3. Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) | |
|---|---|
| by Intensity- Safety Population (N=) | 43 |
| Table 14.3.1.4 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Relationship - Safety Population (N=) | 44 |
| Relationship - Safety Population (N-) | 44 |
| Table 14.3.1.5 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Action taken- Safety Population (N=) | 45 |
| Table 14.3.1.6 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Event Action Taken- Safety Population (N=) | 46 |
| Table 14.3.1.7 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Resolution- Safety Population (N=) | 47 |
| 14.3.2 SERIOUS ADVERSE EVENTS | 49 |
| Table 14.3.2.1 Summary of Overall Serious Adverse Events -Safety Population (N=) | 49 |
| Table 14.3.2.2. Summary of Serious Adverse Events by System Organ Class (SOC) and Preferred Term (PT) -Safety Population (N=) | 51 |
| 14.3.3 CONCOMITANT MEDICATION | 52 |
| Table 14.3.3.1 Summary of Concomitant Medication -Safety Population (N=) | 52 |
| 1.2 LISTINGS | 53 |
| 16.2 PATIENT DATA LISTINGS | 53 |
| Listing 16.2.1 Listing of Patient Study Completion Status | 53 |
| Listing 16.2.2 Listing of Protocol Deviation | 54 |
| Listing 16.2.3 Listing of Informed Consent | 55 |
| Listing 16.2.4 Listing of Inclusion/Exclusion Criteria | 56 |
| 16.2.5 LISTING OF DEMOGRAPHICS | 57 |
| Listing 16.2.5.1 Listing of Demographics at Screening | 57 |
| Listing 16.2.5.2 Listing of Medical History | 58 |
| 16.2.6 LISTING OF SAFETY ANALYSIS | 59 |

# JSS Medical Research India Private Limited Data Management



| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

| Listing 16.2.7.1 Listing of Adverse Event | 59 |
|-----------------------------------------------------------------------|----|
| 16.2.8 LABORATORY TEST | 60 |
| Listing 16.2.8.1 Listing of Coagulation Assessment | 60 |
| Listing 16.2.8.2 Listing of Haematology | 61 |
| Listing 16.2.8.3 Listing of Chemistry | 62 |
| 16.4 INDIVIDUAL PATIENT DATA LISTINGS | 63 |
| Listing 16.4.1 Listing of Treatment Period IMP Dose 1 and Assessments | 63 |
| Listing 16.4.2 Listing of Physical Examination | 64 |
| Listing 16.4.3 Listing of Vital Signs | 65 |
| Listing 16.4.4 Listing of Concomitant Medication | 66 |
| Listing 16.4.5 Listing of Pharmacokinetic Sampling | 67 |

| Cumberland<br>Pharmaceuticals<br>Inc. | JSS Medical Resea<br>Data | red SS RESPONSIVE RELIABLE RESULTS | |
|---|---|---|---|
| Statistical Analysis Plan | | | |
| SOP Number:<br>JSS-DM-BIS-01 | Current Version<br>Number:1.0 | Previous Version Number:<br>None :None | Document<br>Date:06NOV2019 |

## List of Abbreviations and Definition of Terms

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE(s) | Adverse event(s) |
| AUC | Area Under the Curve |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| Cmax | Maximum concentration |
| FDA | Food and Drug Administration |
| IMP | Investigational Medicinal Product |
| IV | Intravenous |
| JSS India | JSS Medical Research India Private Limited |
| kg | Kilogram |
| λ | Terminal elimination rate constant |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mL | Milliliter |
| N | Number of Subjects |
| NSAID | Nonsteroidal anti-inflammatory drug |
| OTC | Over the Counter |
| PEK | Pharmacokinetic-evaluable Population |
| PRN | pro re nata (as necessary) |
| PK | Pharmacokinetics |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TEAE | Treatment-emergent adverse event |
| TLGs | Tables, Listings and Graphs |
| T1/2 | Half-life |
| Tmax | Time to maximum concentration |

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

SOP Number: Current Version Previous Version Number: Document Number: 1.0 None:None Date:06NOV2019

### 1.0 INTRODUCTION

This Statistical Analysis Plan (SAP) describes a comprehensive and detailed description of strategy and statistical technique to be used to realize the analysis of data for Cumberland Pharmaceuticals Inc. protocol CPI-CL-022 (A Multi-Center, Open-Label, Pharmacokinetic, and Safety Study for Reduction in Fever or Management of Pain in Pediatric Subjects Aged Birth to Six Months).

This is a phase 4 study to determine the pharmacokinetics (PK) and safety of single and/or multiple doses of intravenous ibuprofen administered over 10 minutes in children less than six months of age. This study will investigate the application of intravenous ibuprofen in the treatment of pain and/or fever.

The reader of this SAP is encouraged to also read the clinical protocols for details on the conduct of this study and the operational aspects of clinical assessments and timing for completing a patient in this study.

The purpose of this SAP is to outline the planned analyses to be completed to support the completion of the Clinical Study Report (CSR) for protocol CPI-CL-022. The planned analyses identified in this SAP will be included in regulatory submissions and/or future manuscripts. In addition, exploratory analyses not necessarily identified in this SAP may be performed to support the clinical development program. Any post-hoc, or unplanned, analyses which is not identified in this SAP will be clearly identified in the respective CSR.

### 2.0 DESCRIPTION OF THE PROTOCOL

#### 2.1 Protocol Number

CPI-CL-022

#### 2.2 Protocol Title

A Multi-Center, Open-Label Pharmacokinetic and Safety Study for Reduction in Fever or Management of Pain in Pediatric Subjects Aged Birth to Six Months.

#### 2.3 Date

01Jun2015

#### 2.4 Amendment

Amendment 02 dated 30Sep2016

#### 3.0 STUDY OBJECTIVES AND ENDPOINTS

### 3.1 Study Objectives

#### 3.1.1 Primary Objectives

The primary objective of this study is to evaluate the PK profile of a single dose of intravenous ibuprofen administered over approximately 10 minutes.

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

SOP Number: Current Version Previous Version Number: Document Number: 1.0 None :None Date:06NOV2019

#### 3.1.2 Secondary Objectives

The secondary objective of this study is to evaluate the safety of single and repeated doses of intravenous ibuprofen administered to hospitalized pediatric patients by assessing treatment emergent adverse events, vital signs, and laboratory assessments.

#### 3.2 End Points

#### 3.2.1 Primary Pharmacokinetic Endpoints

To evaluate the primary objective of PKs, the following endpoint will be measured:

- Clearance
- Volume of distribution
- Elimination  $T_{1/2}$
- C<sub>max</sub>,
- AUC (0-∞, 0-t)

#### 3.2.2 Secondary (Safety) Endpoints

To evaluate safety, the following endpoints will be measured:

- Treatment emergent adverse events
- Vital signs (temperature, heart rate, respiratory rate, blood pressure)
- Clinical chemistry, hematology, and coagulation assessments

#### 4.0 STUDY METHODS

#### 4.1 Study Design and Plan

This multi-center, open-label, single and/or multiple dose clinical study will assess the PKs (following a single dose) and safety during and after the administration of intravenous ibuprofen. A total of twenty-four subjects, between the ages of birth (> 37 weeks gestational age) to less than six months of age, will be enrolled at up to five clinical centers. The study duration will be up to 72 hours.

This 72-hour study will consist of a Screening/Baseline Period (up to 48 hours prior to the first dose of IMP), a Treatment Period (beginning with the first dose of IMP and continuing for 48 hours) and a Post-Treatment Period (beginning at the end of the Treatment Period and continuing for 24 hours).

The Screening/Baseline Period may begin up to 48 hours prior to Study Hour 0. During the Screening/Baseline Period an evaluation of the inclusion and exclusion criteria, a complete medical history, and a physical examination will be conducted. A review of the subject's pre- IMP vital signs, baseline signs and symptoms, including pain scores (if applicable), concomitant medications, and laboratory assessments will be also conducted to establish the subject's eligibility to participate in the study. The Treatment Period will begin at Hour 0 when an initial dose of investigational medicinal product will be administered over a 10-minute period. Subsequent doses of IMP will be administered, at the investigator's discretion, every 6 to 8 hours, as needed, during the 48-hour treatment period. The total daily dose should not exceed 40 mg/kg/day. Pharmacokinetic sampling will be performed utilizing a sparse sampling technique following the initial dose of IMP. Vital signs, pain scores (if applicable), laboratory assessments and concomitant medications will be monitored during the treatment periods. All treatment emergent adverse events (AEs) will be monitored during the treatment and post-treatment periods. All treatment emergent adverse events will be followed until resolution or stabilization, regardless of the assessment of severity or relationship to the study drug.

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

#### 4.2 Study Initiation and Completion

The study duration will be up to 72 hours and will consist of a Screening/Baseline Period (up to 48 hours prior to the first dose of IMP), a Treatment Period (beginning with the first dose of IMP and continuing for 48 hours) and a Post-Treatment Period (beginning at the end of the Treatment Period and continuing for 24 hours).

#### 4.3 Selection of Study Population

A total of twenty-four subjects, between the ages of birth (> 37 weeks gestational age) to less than six (6) months of age, will receive IMP.

#### **4.3.1** Screening Population (SCREEN)

The Screening Population includes all subjects who provide informed consent and provide demographic and/or baseline screening assessments in the trail.

#### 4.3.2 Safety population

The safety analysis population consists of all participants who were enrolled and received at least part of the IMP; no treated participants will be excluded from the safety analysis population. Safety analysis will be conducted on an as treated basis.

#### 4.3.3 PK (Pharmacokinetics) -evaluable Population

Participants who received the single dose of IMP over the 10-minute infusion period and have the primary PK assessments in the 48hour study period will be eligible for inclusion in the pharmacokinetic-evaluable population (PEP).

#### 4.4 Study Subject Group

There is only subject group: Total of twenty-four subjects, between the ages of birth (> 37 weeks gestational age) to less than six (6) months of age.

#### 4.5 Study Background

Ibuprofen is a nonsteroidal anti-inflammatory drug (NSAID) that was first approved for marketing as a prescription drug in the United States (US) in 1974. Oral ibuprofen is currently approved for use as oral treatment for minimal to moderate pain from arthritis, surgery, sunburn, menstruation, and fever. Like aspirin and other drugs in the NSAID family, ibuprofen is believed to reduce the inflammatory response by inhibiting the formation of prostaglandins.

CALDOLOR® (ibuprofen) Injection was approved by the US Food and Drug Administration in June 2009 for adults and in May 2016 for pediatric patient greater than six months of age. CALDOLOR is indicated in adults and pediatric patients 6 months and older for the management of mild to moderate pain, management of moderate to severe pain as an adjunct to opioid analgesics and for the reduction of fever. This formulation of intravenous (IV) ibuprofen is now being studied for use in the pediatric population less than 6 months of age.

#### 4.6 Study Rationale

For the pediatric patient population, there are multiple oral over-the-counter (OTC) ibuprofen products available for the treatment of pain in children. Motrin® (McNeil Consumer Healthcare, Fort

Protocol No. CPI-CL-022 Confidential 06Nov2019
Statistical Analysis Plan 

# JSS Medical Research India Private Limited Data Management



## Statistical Analysis Plan

SOP Number: Current Version Previous Version Number: Document Number: 1.0 None: None Date:06NOV2019

Washington, Pennsylvania) is one of the most commonly used oral ibuprofen products currently marketed. The recommended dose for Motrin for treatment of pain in children 6 months to 12 years of age is 10 mg/kg with the recommended maximum daily dose of 40 mg/kg. The recommended dosing for children 12 years of age and older is the same as that used for adults, 200 to 800 mg up to four times daily, with a maximum of 3200 mg per day whereas the population for this study will consist of hospitalized pediatric subjects from birth (> 37 weeks gestational age) to < 6 months of age with a clinical indication of pain and/or fever.

#### 4.7 Schedule of Study Events

There will be three scheduled visits in the study. For an example:

Visit 1: Screening/Baseline (up to 48 hours prior to the first dose of IMP)

Visit 2: Treatment Period (beginning with the first dose of IMP and continuing for 48 hours)

Visit 3: Post-Treatment Period (beginning at the end of the Treatment Period and continuing for 24 hours)

#### 4.8 Schedule of Visits and Procedures

Schedule of visits is shown in Table 4.8

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

Table 4.8 Overall schedule of time and events

| | Study Period | | | |
|---|---|---|---|---|
| Measurement/Evaluation | Screening/<br>Baseline | Treatment | | Post-<br>Treatment |
| Time(s) | Hour - 48 to<br>Hour 0 | Hour 0 to Hour<br>24 | Hour 24 to<br>Hour 48 | Hour 48 to<br>Hour 72 |
| Informed Consent | X | | | |
| Inclusion/Exclusion Criteria | X | | | |
| Medical History | X | | | |
| Physical Examination | X | | | |
| Demographic Data | X | | | |
| Baseline Signs & Symptoms | X | | | |
| Vital Signs | X | X | X | XΨ |
| Laboratory Assessments | X+ | X: | | XΨ |
| Pharmacokinetic Assessments | | $X^{\phi}$ | | |
| Concomitant Medications | X <sup>+</sup> | X | X | |
| IMP Administration (Initial & PRN) | | X | X | |
| Adverse Event Monitoring | | X** | X** | X** |

IMP = Investigational Medicinal Product

\*Laboratory Assessment and Vital Signs must be performed at Study Hour 72 (± 6 hours) or at the time of discharge, whichever occur first.

### 5.0 GENERAL CONSIDERATIONS FOR STATISTICAL ANALYSIS

#### 5.1 Sample Size Determination

A total of 24 subjects will be enrolled in the study. No power calculations will be performed.

#### 5.2 Method of Treatment Assignment and Randomization

All subjects who meet all the inclusion and exclusion criteria during the Screening/Baseline Period will be enrolled into the study. Only eligible subjects will be assigned to receive intravenous ibuprofen, 10 mg/kg per dose. There is no randomization; this study is open-label with respect to the treatment assignment.

#### 5.3 Methods for Withdrawals and Missing Data

If the subject is withdrawn from the study, data collected on the subject up to the time of withdrawal must remain in the trial database (FDA 2008).

Statistical Analysis Plan 

<sup>\*</sup>Laboratory data collected within 48 hours prior to dosing may be used for Screening/Baseline Period laboratory assessments.

<sup>&</sup>lt;sup>+</sup> Record concomitant medication actually administered to the subject in the 8 hours prior to the first dose of IMP. <sup>φ</sup> PK assessment must be taken immediately following the first dose of IMP then per the sparse sampling schedule. <sup>s</sup> Laboratory Assessment must be performed at Study Hour 24 (± 6 hours)

<sup>\*\*</sup>All treatment adverse events will be followed until resolution or stabilization, regardless of the assessment of severity or relationship to the study drug.

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

SOP Number: Current Version Previous Version Number: Document Number: 1.0 None:None Date:06NOV2019

If a decision is made to withdraw the subject from the study; the investigator should clarify with the subject's parent or legal guardian if the subject is to be withdrawn from all components of the study or if the subject is withdrawn from the primary interventional component but if the subject's parent or legal guardian would be willing to allow the investigator to continue other research activities as described below and in the informed consent:

- Medical course or laboratory results obtained through non-invasive chart review
- Vital signs, as outlined in the protocol
- Adverse event monitoring, as outlined in the protocol
- Post-Treatment follow-up

If required, subjects will be replaced to ensure a total of 24 PK-evaluable subjects. The replacement criteria are given below.

Subjects who are enrolled into the study but do not receive any IMP will be replaced. Subjects who withdraw from the study after receiving IMP but who do not complete the PK portion of the study within the first 4 hours will also be replaced.

No statistical imputation will be incorporated for the missing values.

### 5.4 Analysis Software

All analysis will be performed using SAS® Software version 9.4 or later.

#### 6.0 DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

#### 6.1 Demographics

During the Screening/Baseline Period, the Demographic date (age, race, ethnicity, height, weight) will be captured and analyzed using descriptive statistics (mean, median, standard deviation (SD), minimum and maximum) for continuous variables and using frequency count and percentage for categorical variables.

#### 6.2 Baseline and Screening Conditions

Descriptive statistics (mean, median, standard deviation (SD), minimum and maximum) for continuous variables and frequency count and percentage for categorical variables will be presented for all baseline characteristics such as physical examination, vital signs and laboratory parameters.

During the Screening/Baseline Period, the following evaluations will be performed to determine the subject's eligibility for this study:

- Informed consent (by parent or legal guardian)
- Inclusion and exclusion criteria
- Complete medical history
- Physical examination
- Demographic date (age, race, ethnicity, weight, sex)
- Baseline signs & symptoms
- Vital signs (temperature, heart rate, respiratory rate, and blood pressure)
- · Laboratory assessment
- · Concomitant medications


#### Cumberland JSS Medical Research India Private Limited RESPONSIVE **Pharmaceuticals** RELIABLE **Data Management** RESULTS Inc. Statistical Analysis Plan SOP Number:

#### 6.3. **Baseline Medical History**

JSS-DM-BIS-01

Current Version

Number: 1.0

The medical history should be recorded at Screening/Baseline and should include history of hepatic, renal, neurological, endocrine, cardiovascular, and pulmonary disease, operations, serious illnesses and any other condition the investigator feels is significant. Medical history should include information related to the duration, i.e. the number of months must be recorded in the case report form. Subjects reporting Medical History will be presented by using frequency (percentage) count.

None:None

Previous Version Number:

Document

Date:06NOV2019

#### 6.4 **Physical Examination**

Frequency count (percentage) of subjects will be presented for each Body System.

#### 7.0 STATISTICAL ANALYSES

The primary objective of this study is to evaluate the PK profile of a single dose of intravenous ibuprofen administered over approximately 10 minutes.

#### 7.1 **Primary Endpoint Analysis (Pharmacokinetic Parameters)**

PK samples will be collected on all subjects immediately (± 5 minutes) following completion of the first dose of intravenous ibuprofen; then alternating subjects will have PK sampling performed at 30 minutes and 2 hours or at 1 hour and 4 hours following the first dose of intravenous ibuprofen (12 subjects will have samples collected immediately following the first dose, then at 30 minutes and 2 hours; and, 12 subjects will have samples collected immediately following the first dose, then at 1 hour and 4 hours). Pharmacokinetic sampling will only be performed following the first dose of IMP regardless of the total number of doses of IMP administered.

To evaluate the PKs, the following parameters will be measured:

- Clearance
- Volume of distribution
- Elimination T<sub>1/2</sub>
- $C_{\text{max}}$
- $AUC(0-\infty, 0-t)$

On the basis of plasma ibuprofen concentration time data, the following PK parameters will be estimated by using a non-compartmental model:

- AUC<sub>0-t</sub>, calculated by using the linear-log trapezoidal rule: linear trapezoidal rule up to time to maximum concentration, and then a log trapezoidal rule for the remainder of the curve, where t corresponds to the last measurable time point
- $AUC_{0-\infty} = AUC_{0-t} + C_t/\lambda_z$ , where  $C_t$  is the last measurable ibuprofen concentration and  $\lambda_z$  is the terminal elimination rate constant calculated by using log linear regression of the terminal elimination phase of the plasma concentration versus time curve
- C<sub>max</sub> of ibuprofen estimated by inspection of the ibuprofen concentration time curve
- T<sub>max</sub> estimated by inspection of the ibuprofen concentration time curve
- Terminal  $T_{1/2} = \ln (2)/\lambda_z$
- Clearance=Renal Blood Flow\* extraction ratio
- Volume of distribution= Clearance/  $\lambda_z$

#### 7.2 **Secondary Endpoint Analysis**

# JSS Medical Research India Private Limited Data Management



### Statistical Analysis Plan

| SOP Number: | Current Version | Previous Version Number: | Document |
|---------------|-----------------|--------------------------|----------------|
| JSS-DM-BIS-01 | Number:1.0 | None :None | Date:06NOV2019 |

The secondary objective of this study is to evaluate the safety of single and repeated doses of intravenous ibuprofen administered to hospitalized pediatric patients by assessing treatment emergent adverse events, vital signs, and laboratory assessments. The participant population of interest for the safety analyses is the safety analysis population.

Safety will be evaluated on the basis of treatment emergent AEs. AE data will be listed individually and summarized by body system organ class and preferred terms within system organ class (MedDRA). Serious and/or unexpected AEs will also be discussed on a case by case basis. Each AE will be counted only once for a given participant. If the same AE occurs on multiple occasions, the highest severity and least favorable relationship reported will be assumed. If two or more AEs are reported as a unit, the individual terms will be reported as separate experiences.

#### 8.0 SAFETY AND TOLERABILITY ANALYSES

The analysis of safety assessments in this study will include summaries of the following categories of safety and tolerability data collected for each subject:

- Adverse Events
- Physical examination
- Vital Signs
- > Concomitant Medication
- Laboratory Parameters

#### **8.1** Adverse Events

Adverse events will be assessed regularly during the Treatment Period. Adverse event collection will begin at the start of IMP administration and continue through Study Hour 48 or discharge, whichever comes first. Subjects do not need to remain hospitalized for the 48-hour Treatment Period. All treatment emergent adverse events will be monitored until resolution or stabilization, regardless of the assessment of severity or relationship to the study drug. All AEs, observed by, documented in the subject's medical record, or reported to the research team must be recorded in both the subject's research record and the case report form.

#### 8.2 Vital Signs

Descriptive statistics will be presented for each test at baseline, treatment period and post-treatment period.

#### 8.3 Concomitant Medication

Concomitant medications, during the study will be listed by subject and summarized for the enrolled population as counts and percentage.

### 8.4 Laboratory parameters

The summary of following laboratory parameters will be provided through descriptive statistics:

- o Sodium
- o Potassium

#### Cumberland JSS Medical Research India Private Limited RESPONSIVE **Pharmaceuticals** RELIABLE **Data Management** RESULTS Inc. **Statistical Analysis Plan** SOP Number: Current Version Previous Version Number: Document Number: 1.0 None:None Date:06NOV2019 JSS-DM-BIS-01

- o Chloride
- o Total carbon dioxide
- o Glucose
- o Blood urea nitrogen
- Creatinine
- Total bilirubin
- o Albumin
- o Total protein
- Aspartate aminotransferase
- Alanine aminotransferase
- Lactate dehydrogenase
- Hematology and coagulation include:
- White blood cellcount and differential
- Hematocrit
- Hemoglobin
- Platelets
- o Prothrombin time
- o Partial thromboplastin time

### 9.0 INTERIM ANALYSIS OR OTHER PLANNED ANALYSES

No interim analysis is planned in this study.

#### 10.0 REPORTING CONVENTIONS

#### 10.1 Reporting of Numeric Values

All raw data will be presented to the original number of decimal places. The mean, median and quartiles will be presented with 1 decimal place more than raw data. The standard deviation (SD), Standard Error of Mean and Confidence Interval (CI) of mean will be presented with 1 decimal place more than mean. The range (minimum and maximum) will be presented as per the raw data Percentages will be presented in xx.x% format. All categories of variables will be presented even if there is no data. Blank cells will be filled by "-"in reporting of results.

Precision of p-values will be 4 decimal places. p-values less than 0.0001 will be presented as <0.0001 and if equal to 1 then  $\ge 0.9999$ 

### 11.0 Output (Tables, Listings and Graphs) Considerations

The default Tables, Listings and Graphs (TLG) layout will be as follows.

| Orientation | All pages should preferably be landscape. |
|-------------|-------------------------------------------|
| Paper Size | Legal size |
| Margins | Top: 1 in Bottom: 0.75 in Left: 0.75 in |

#### Cumberland JSS Medical Research India Private Limited RESPONSIVE **Pharmaceuticals** RELIABLE **Data Management** RESULTS Inc. Statistical Analysis Plan SOP Number: Current Version Previous Version Number: Document Number: 1.0 None:None Date:06NOV2019 JSS-DM-BIS-01

| | Right: 0.75 in |
|---------|-------------------------------------------------|
| Font | Font style (preferably Courier New) of the Text |
| | Titles of Table/Listing will be center |
| | Left |
| Headers | Sponsor: |
| | Study Name: |
| | Protocol No: |
| | Left |
| | Analyst Initials: |
| | Program Name: |
| Footers | Program Run date: time: |
| | Right |
| | Datasets Used: |
| | Page XXX of YYY |

The margin may be reduced as necessary to allow additional rows to be presented, but not at the expense of clarity. In addition, the orientation may be changed to portrait if appropriate. The date format for all presentations will be 'DDMMMYYYY'.

#### 12.0 REFERENCES

- 1. Protocol: CL022 Amendment02 30SEP2016 FINAL
- 2. Case Report Form (CRF), CRF CL022\_Amendment02\_30SEP2016\_FINAL.
- 3. ICH E3: Structure and content of Clinical Study Reports, November 1995, CPMP.
- 4. ICH E9: Statistical Principles for Clinical Trials, September 1998, CPMP

#### 

### **APPENDIX 1: SUMMARY OF STATISTICAL ANALYSIS**

### 1.1 TABLES

### 14.1.1 Subject Disposition

#### Table 14.1.1.1 Summary of Inclusion/Exclusion Criteria – All Screened (N=)

All Screened (N=)

Inclusion/Exclusion Criteria, n (%) [1]

Number of Subjects meeting all Inclusion Criteria

Number of Subjects meeting at least one exclusion criteria

Number of eligible subjects

Number of Subjects Screened

Source: Listing 16.2.4

Note

[1] Percentage will be calculated by taking respective column header count as denominator.

## JSS Medical Research India Private Limited **Data Management**



### Title: Statistical Analysis Plan

SOP Number: Current Version Number 1.0 Previous Version Number:None Document Date:06NOV2019 JSS-DM-BIS-01

Table 14.1.1.2 Summary of Study Populations – All Enrolled (N=)

Category, n (%) [1]

Overall (N=)

Screened Population

No. of Subjects in Safety Population

No. of Subjects Completed Study

No. of Subjects Discontinued study

Reason for pre-mature discontinuation [2]

Subject withdrew from the study /Consent withdrawn

The investigator withdrew the subject from the study

The subject was discontinued from the study secondary to an AE

or SAE

Subject non-compliance

**Enrollment Violation** 

Excluded medication, Procedure, or Therapy

Other reason

**Source:** Listing 16.2.1 and Listing 16.2.3

[1] Percentage will be calculated taking respective column header group count as denominator.

[2] Percentage will be calculated using total number of discontinued subjects count as denominator.

| Cumberland |
|----------------------|
| Pharmaceuticals Inc. |

## **JSS Medical Research India Private Limited Data Management**



# **Title: Statistical Analysis Plan**

| | | <u> </u> | |
|---|---|---|---|
| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

### 14.1.2 Demographics and Baseline Characteristics

Table 14.1.2.1 Summary of Subject Demographics-Safety Population (N=)

| Parameters | Statistic/Category, n (%) [1] | Overall (N=) |
|---|---|---|
| Gender | | |
| | Male | |
| | Female | |
| Age (in days) | | |
| | n | |
| | Mean | |
| | SD | |
| | Median | |
| | Range (Min: Max) | |
| Race | | |
| | American Indian or Alaskan Native | |
| | Asian | |
| | Black or African American | |
| | Native Hawaiian or other Pacific Islander | |
| | White | |
| | Multi-racial | |
| | Other | |
| Ethnicity | Otilci | |
| Etimenty | Hispanic or Latino | |
| | Non-Hispanic or Non-Latino | |
| Height (cm) | Non-mispaine of Non-Latino | |
| Height (Chi) | , | |
| | n<br>Maria | |
| | Mean | |
| | SD | |
| | Median | |
| W. ' 1 (IZ ) | Range (Min: Max) | |
| Weight (Kg) | | |
| | n | |
| | Comitation | 001.0.2019 |

# JSS Medical Research India Private Limited Data Management



| Title: | <b>Statistical</b> | <b>Analysis</b> | Plan |
|--------|--------------------|-----------------|------|
|--------|--------------------|-----------------|------|

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0

Previous Version Number:None

Document Date:06NOV2019

Mean SD Median Range (Min:Max)

Source: Listing 16.2.5.1

Note:

[1] Percentage will be calculated taking respective column header group count as denominator.

General Note:

Days=month\*30.42

# JSS Medical Research India Private Limited Data Management



## Title: Statistical Analysis Plan

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0


Document Date:06NOV2019

### 14.1.3 Medical History

Table 14.1.3.1 Summary of Medical History by SOC and PT-Safety Population (N=)

| System Organ Class | Preferred Term, n (%) [1] | Overall(N=) |
|----------------------|---------------------------|-------------|
| Total (All SOC/PT) | Any | |
| System Organ Class 1 | Any | |
| | Preferred term1 | |
| | Preferred term2 | |
| System Organ Class 2 | Any | |
| | Preferred term1 | |
| | Preferred term2 | |

**Source Data:** Listing 16.2.5.2

Note:

[1] Percentages will be calculated by taking respective column header group count as denominator.

#### General Note:

- Medical History will be coded using MedDRA version 21.1 or later.
- NA: Not Applicable

# JSS Medical Research India Private Limited Data Management



## Title: Statistical Analysis Plan

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0


Document Date:06NOV2019

### 14.1.4 Physical Examination

Table 14.1.4.1 Summary of Physical Examination--Safety Population (N=)

| Parameters | Statistic/Category, n (%) [1] | Overall (N=) |
|---|---|---|
| Was Physical examination done? [1] | | |
| | Yes | |
| | No | |
| General Appearance, [2] | | |
| | Normal | |
| | Abnormal | |
| | Not Assessed | |
| HEENT | | |
| | Normal | |
| | Abnormal | |
| | Not Assessed | |
| Cardiovascular | | |
| | Normal | |
| | Abnormal | |
| | Not Assessed | |
| Respiratory | | |
| • | Normal | |
| | Abnormal | |
| | Not Assessed | |

**Source Data:** Listing 16.4.2

Note

#### **Programming Note:**

The same table will be repeated for all the available visits and all the physical examination – Gastrointestinal, Hepatic, Renal, Genitourinary, Musculokeletal, Endocrine, Immune/Allegry, Central Nervous System, Dermatological, Other.


<sup>[1]</sup> Respective column header group counts will be used as denominator for percentage calculation.

<sup>[2]</sup> Percentages for Physical Examination will be calculated using respected 'Yes' count as denominator.

# JSS Medical Research India Private Limited Data Management



## Title: Statistical Analysis Plan

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0


Document Date:06NOV2019

### 14.2 Efficacy Analysis

### 14.2.1 Primary Efficacy Analysis

Table 14.2.1.1 Summary of Statistics of Pharmacokinetics (PK) Parameters-PK Population(N=)

| Parameters | Statistic | Overall(N=) |
|------------------------|------------------------------|-------------|
| Clearance | | |
| | n | |
| | Mean | |
| | Geometric Mean | |
| | Standard Deviation | |
| | Median | |
| | Coefficient of Variation (%) | |
| | Range (Min.:Max.) | |
| Volume of distribution | | |
| | n | |
| | Mean | |
| | Geometric Mean | |
| | Standard Deviation | |
| | Median | |
| | Coefficient of Variation (%) | |
| | Range (Min.:Max.) | |

Protocol No. CPI-CL-022 Statistical Analysis Plan Confidential

06Nov2019

# JSS Medical Research India Private Limited Data Management



## **Title: Statistical Analysis Plan**

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0


Document Date:06NOV2019

Elimination T1/2

n

Mean

Geometric Mean

Standard Deviation

Median

Coefficient of Variation (%)

Range (Min.:Max.)

Cmax

n

Mean

Geometric Mean

Standard Deviation

Median

Coefficient of Variation (%)

Range (Min.:Max.)

Tmax

n

Mean

Geometric Mean

Standard Deviation

# JSS Medical Research India Private Limited Data Management



| Title: | <b>Statistical</b> | <b>Analysis</b> | Plan |
|--------|--------------------|-----------------|------|
|--------|--------------------|-----------------|------|

SOP Number: JSS-DM-BIS-01

Current Version Number 1.0


Document Date:06NOV2019

Median

Coefficient of Variation (%)

Range (Min.:Max.)

 $AUC(0-\infty, 0-t)$ 

n

Mean

Geometric Mean

Standard Deviation

Median

Coefficient of Variation (%)

Range (Min.:Max.)

#### Note

[1] Any observation with concentration value of 0.000 will be ignored while deriving the geometric mean. General Note:

• Any concentration below this limit of quantification is reported as 0.000.

# JSS Medical Research India Private Limited Data Management



# **Title: Statistical Analysis Plan**

SOP Number: JSS-DM-BIS-01

Current Version Number 1.0


Document Date:06NOV2019

### 14.2.2 Secondary Analysis (Safety Endpoint)

### Table 14.2.2.1 Summary of Overall Treatment Emergent Adverse Events -Safety Population (N=)

| | | Events (N | (N=) Patients (N=) | % of Patien |
|---|---|---|---|---|
| Category | Parameter, n (%) [1] | 2,0110 (1 | 1 40101105 (11) | 70 01 1 40101 |
| TOTAL<br>Serious Adverse Events | | | | |
| Serious Adverse Events | Yes | | | |
| | No | | | |
| Intensity | | | | |
| | Mild | | | |
| | Moderate | | | |
| | Serve | | | |
| Resolution | | | | |
| | Resolved | | | |
| | Resolved with Sequelae | | | |
| | Chronic condition | | | |
| | Fatal | | | |
| | Unknown | | | |
| IMP Action Taken | | | | |
| | None | | | |
| | IMP Interrupted | | | |
| | IMP Discontinued | | | |

# JSS Medical Research India Private Limited Data Management



## **Title: Statistical Analysis Plan**

| CODN 1 | | | |
|---|---|---|---|
| SOP Number: | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
| JSS-DM-BIS-01 | Current version runnoerr. | Trevious version runnoer.runne | Bocument Bate.00110 v 2017 |

| | | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|
| Category | Parameter, n (%) [1] | , , | | |
| Event Action taken | | | | |
| | None | | | |
| | Concomitant Medication | | | |
| | Hospitalization (complete SAE) | | | |
| | Other | | | |
| Relationship of the event to | | | | |
| the IMP | | | | |
| | Not Related | | | |
| | Possibly Related | | | |
| | Related | | | |

**Source Data: Listing** 16.2.7.1

#### Note

[1] Percentages will be calculated using respective column header counts as denominator.

#### General Note

• Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.

# JSS Medical Research India Private Limited Data Management



## Title: Statistical Analysis Plan

| | | v | |
|---|---|---|---|
| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

Table 14.2.2.2. Summary of Treatment Emergent Adverse Events by System Organ Class (SOC) and Preferred Term (PT)- Safety Population (N=)

| Preferred Term, | | | |
|---|---|---|---|
| n(%) [1] | Events (N=) | Patients (N=) | % of Patients |
| NA | | | |
| ANY | | | |
| PT1 | | | |
| PT2 | | | |
| ANY | | | |
| PT1 | | | |
| PT2 | | | |
| | NA ANY PT1 PT2 ANY PT1 | NA ANY PT1 PT2 ANY PT1 | NA ANY PT1 PT2 ANY PT1 |

Source Data: Listing 16.2.7.1

#### Note:

[1] Percentages will be calculated using respective column header counts as denominator.

NA: Not Applicable.

#### **General Note:**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 [0] (0.0%) ".

## **JSS Medical Research India Private Limited Data Management**



# **Title: Statistical Analysis Plan**

| SOP Number: | | | |
|---|---|---|---|
| JSS-DM-BIS-01 | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |

Table 14.2.2.3 Summary of Vital Signs – Safety Population (N=)

| Parameters | Statistic/Category, n (%) [1] | | V | isit | |
|---|---|---|---|---|---|
| | | Screening | Treatment<br>Period<br>(0-24 hours) | Treatment<br>Period<br>(24-48 hours) | Post-<br>Treatment<br>Period |
| Temperature | | | | , | |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Heart Rate | | | | | |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Respiratory Rate | Tange (Trans Trans) | | | | |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Systolic Blood Pressu | re | | | | |
| • | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Diastolic Blood | | | | | |
| Pressure | | | | | |
| | n | | | | |
| Protocol No. CPI-CL | -022 | Confidentia | a1 | | 06Nov2019 |

# JSS Medical Research India Private Limited Data Management



| Title: | <b>Statistical</b> | <b>Analysis</b> | Plan |
|--------|--------------------|-----------------|------|
|--------|--------------------|-----------------|------|

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0


Document Date:06NOV2019

Mean SD

Median

Range (Min: Max)

**Source Data:** Listing 16.4.3

Note:

[1] Respective column header group counts will be used as denominator for percentage calculation.

# JSS Medical Research India Private Limited Data Management



# **Title: Statistical Analysis Plan**

|---|---|---|---|
| JSS-DM-BIS-01 | Current version runneers. | Trevious version runnervone | Bocament Bate:00110 12017 |

Table 14.2.2.4 Summary of Coagulation Assessments – Safety Population (N=)

| | | Visit | | | |
|---|---|---|---|---|---|
| | Statistic/Category, n<br>(%) [1] | Screening/Baselin<br>e Study Hour -48<br>to<br>Hour 0) | Treatment Period<br>(Study Hour 0 to<br>Hour<br>24) +/- 6 hrs | Treatment Period (Study<br>Hour 24 to<br>Hour 48) +/- 6 hrs | Post-Treatment Period (Study Hour 48 to Hour 72) +/- 6 hrs |
| Prothrombin time (PT) | | , | , | | , |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Clinically Significant | | | | | |
| | Yes | | | | |
| | No | | | | |
| Activated Partial | | | | | |
| Thromboplastin Time (aPTT) | | | | | |
| • | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Clinically Significant | | | | | |
| , , | Yes | | | | |
| | No | | | | |
| International Normalized | | | | | |
| Ratio (INR) | | | | | |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |

# JSS Medical Research India Private Limited Data Management



| Title: | <b>Statistical</b> | <b>Analysis</b> | Plan |
|--------|--------------------|-----------------|------|
|--------|--------------------|-----------------|------|

| SOP Number: | Compant Warrian Number 1 0 | Dunious Vagaina Naughau Naug | Decompost Detail (NOV2010 |
|---|---|---|---|
| JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

Clinically Significant

Yes

No

Source Data: Listing 16.2.8.1

Note

[1] Respective column header group counts will be used as denominator for percentage calculation.

## **JSS Medical Research India Private Limited Data Management**



# **Title: Statistical Analysis Plan**

| SOP Number: | | | |
|---|---|---|---|
| | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
| JSS-DM-BIS-01 | | | 200000000000000000000000000000000000000 |

Table 14.2.2.5 Summary of Haematology – Safety Population (N=)

| | | Visit | | | |
|---|---|---|---|---|---|
| Parameters | Statistic/Category, n (%) [1] | Screening/Baseline<br>Study Hour -48 to<br>Hour 0) | Treatment Period (Study<br>Hour 0 to Hour<br>24) +/- 6 hrs | Treatment Period<br>(Study Hour 24 to<br>Hour 48) +/- 6 hrs | Post-Treatment Period<br>(Study Hour 48<br>to Hour 72) +/- 6 hrs |
| Hemoglobin | | , | , | • | , |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Clinically Significant | | | | | |
| | Yes | | | | |
| | No | | | | |
| Hematocrit | | | | | |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Clinically Significant | | | | | |
| | Yes | | | | |
| | No | | | | |
| Platelets | | | | | |
| | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Range (Min: Max) | | | | |
| Clinically Significant | | | | | |
| | Yes | | | | |
| | No | | | | |
| White Blood Cell Count | | | | | |
| | n | | | | |
#### JSS Medical Research India Private Limited **Data Management**



#### **Title: Statistical Analysis Plan**

| SOP Number: | | D : W : N 1 N | D 4 D 4 00101/2010 |
|---|---|---|---|
| JSS-DM-BIS-01 | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |

Mean SD

Median Range (Min: Max)

Clinically Significant

Yes

No

Total Neutrophil Count (segmented neutrophils plus

bands)

n Mean SD Median

Range (Min: Max)

Clinically Significant

Yes

No

Source Data: Listing 16.2.8.2

[1] Respective column header group counts will be used as denominator for percentage calculation.

**Programming Note:** 

The same table will be repeated for all available Hematology Parameters-Lymphocytes, Monocytes, Eosinophils, Basophils.

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number: | | | |
|---|---|---|---|
| 5 01 1 (01110 41) | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
| JSS-DM-BIS-01 | Carrent version realisers. | Trevious version runneer, rune | Boedinent Bate: 00110 12019 |

Table 14.2.2.6 Summary of Chemistry – Safety Population (N=)

| Parameters Statistic/Category, n (%) [1] Screening/Baseline Study Hour -48 to Hour 0) Study Hour 0 to Hour (Study Hour 24 to Hour 48) +/- 6 hrs Sodium N Mean SD Median Range (Min: Max) Clinically Significant Yes No Potassium N Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate N Mean SD Median Range Mean SD Median Range Mean SD Mo Median Range (Min: Max) Mean SD Median Mean SD Median Mean SD Median Mean SD Median Mean SD Median Mean SD Median Mean SD Median | |
|---|---|
| Sodium Nean SD Median Range (Min: Max) Clinically Significant Yes No No Nedian SD Median Range (Min: Max) Potassium Nean SD Median Range (Min: Max) Clinically Significant Yes No No No No No No No N | Post-Treatment Period (Study Hou<br>48<br>to Hour 72) +/- 6 hrs |
| Mean SD Median Range (Min: Max) Clinically Significant Yes No Potassium In Mean SD Median Range (Min: Max) Clinically Significant Ves No Total Carbon Dioxide/Bicarbonate In Mean SD No Total Carbon Dioxide/Bicarbonate In Mean SD No Total Carbon Dioxide/Bicarbonate | |
| SD Median Range (Min: Max) Clinically Significant Yes No Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD Mean SD Median Range (Min: Max) | |
| Median Range (Min: Max) Clinically Significant Yes No Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD Mean SD Mean SD | |
| Range (Min: Max) Clinically Significant Yes No Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD Mean SD SD No SD | |
| Clinically Significant Yes No Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD Mean SD SD | |
| Clinically Significant Yes No Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD N Mean SD | |
| Yes No Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Potassium n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| n Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Mean SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| SD Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Median Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Range (Min: Max) Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Clinically Significant Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Yes No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| No Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Total Carbon Dioxide/Bicarbonate n Mean SD | |
| Dioxide/Bicarbonate n Mean SD | |
| n<br>Mean<br>SD | |
| Mean<br>SD | |
| Mean<br>SD | |
| SD | |
| Range (Min: Max) | |
| Clinically Significant | |
| Yes | |
| No | |

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

| CODN: 1 | | | |
|---|---|---|---|
| SOP Number: | C | D ' 17 ' N 1 N | D |
| JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

Chloride

n

Mean SD Median

Range (Min: Max)

Clinically Significant

Yes

No

Glucose

n Mean SD Median

Range (Min: Max)

Clinically Significant

Yes

No

Source Data: Listing 16.2.8.3

Note:

[1] Respective column header group counts will be used as denominator for percentage calculation.

#### **Programming Note:**

The same table will be repeated for all the available Chemistry Parameters- Blood Urea Nitrogen, Creatinine, Total Bilirubin, Albumin, Total Protein, Aspartate Transaminase, Alanine Transaminase, Lactate Dehydrogenase

| Cumberland<br>Pharmaceuticals Inc. | earch India Private Limited<br>a Management | RESPONSIVE RELIABLE RESULTS |
|---|---|---|
| Title: Statistical Analysis Plan | | |
| SOP Number: JSS-DM-BIS-01 Current Version Number1.0 Previous Version Number:None Document Date:06NOV2019 | | |

#### **Safety Analysis** 14.3

#### 14.3.1 ADVERSE EVENTS

Table 14.3.1.1 Summary of Overall Adverse Events -Safety Population (N=)

| | | Events ( | N=) Patient | s (N=) % of Patients |
|---|---|---|---|---|
| Category | Parameter, n (%) [1] | 2.0.00 | 2 | 70 011 4000000 |
| TOTAL<br>Serious Adverse Events | | | | |
| | Yes | | | |
| | No | | | |
| Intensity | | | | |
| | Mild | | | |
| | Moderate | | | |
| | Serve | | | |
| Resolution | | | | |
| | Resolved | | | |
| | Resolved with Sequelae | | | |
| | Chronic condition | | | |
| | Fatal | | | |
| | Unknown | | | |
| IMP Action Taken | | | | |
| | None | | | |
| | IMP Interrupted | | | |
| Statistical Analysis Plan | | | | |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number: | | | |
|---|---|---|---|
| SOI I (GIII) OI. | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
| JSS-DM-BIS-01 | Carrent version reamour. | Trevious version runneer, rune | Bocament Bate:00110 12019 |

| | | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|
| Category | Parameter, n (%) [1] | | | |
| | IMP Discontinued | | | |
| Event Action taken | | | | |
| | None | | | |
| | Concomitant Medication | | | |
| | Hospitalization (complete SAE) | | | |
| | Other | | | |
| Relationship of the event to the IMP | | | | |
| | Not Related | | | |
| | Possibly Related | | | |
| | Related | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator.

#### **General Note**

• Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

| | | • | |
|---|---|---|---|
| SOP Number: | Current Version Number 1.0 | Previous Version Number: None | Document Date:06NOV2019 |
| JSS-DM-BIS-01 | Current version Number 1.0 | 1 Tevious version Number. None | Document Date.00110 V 2019 |

Table 14.3.1.2. Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) -Safety Population(N=)

| System Organ Class | Preferred Term, n(%) [1] | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | |
| SOC 1 | ANY | | | |
| | PT1 | | | |
| | PT2 | | | |
| SOC 2 | ANY | | | |
| | PT1 | | | |
| | PT2 | | | |

Source Data: Listing 16.2.7.1

Note

[1] Percentages will be calculated using respective column header counts as denominator.

NA: Not Applicable.

#### **Genral Note:**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

| | | · · | |
|---|---|---|---|
| JSS-DM-BIS-01 | Current version Number 1.0 | 1 Tevious version Number None | Document Date:00NO v 2019 |

Table 14.3.1.3. Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Intensity- Safety Population (N=)

| System Organ Class | Preferred Term, n (%) [1] | Intensity | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | | |
| SOC 1 | ANY | | | | |
| | PT1 | | | | |
| | | Mild<br>Moderate | | | |
| | | Severe | | | |
| | PT2 | | | | |
| | | Mild<br>Moderate | | | |
| | | Severe | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator. General Note

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events] will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

| | | · · | |
|---|---|---|---|
| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

Table 14.3.1.4 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Relationship - Safety Population (N=)

| System Organ Class | Preferred Term | Causality | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | | |
| SOC 1 | ANY | | | | |
| | PT1 | | | | |
| | | Not related | | | |
| | | Possibly Related | | | |
| | | Related | | | |
| | PT2 | | | | |
| | | Not related | | | |
| | | Possibly Related | | | |
| | | Related | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator.

#### **General Note:**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events] will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

| | | · · | |
|---|---|---|---|
| JSS-DM-BIS-01 | Current version Number 1.0 | 1 Tevious version runnoer, runne | Document Date.00110 v 2019 |

Table 14.3.1.5 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Action taken- Safety Population (N=)

| System Organ Class | Preferred Term | Action taken | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | | |
| SOC 1 | ANY<br>PT1 | | | | |
| | | None | | | |
| | | IMP Interrupted | | | |
| | | IMP Discontinued | | | |
| | PT2 | | | | |
| | | None | | | |
| | | IMP Interrupted | | | |
| | | IMP Discontinued | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator.

#### **General Note**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events] will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |
|---|---|---|---|

Table 14.3.1.6 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Event Action Taken- Safety Population (N=)

| System Organ Class | Preferred Term | Outcome | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | | |
| SOC 1 | ANY | | | | |
| | PT1 | | | | |
| | | None | | | |
| | | Concomitant Medication | | | |
| | | Hospitalization | | | |
| | | Other | | | |
| | PT2 | | | | |
| | | None | | | |
| | | Concomitant Medication | | | |
| | | Hospitalization | | | |
| | | Other | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator.

#### **General Note:**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events] will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

Protocol No. CPI-CL-022 Confidential
Statistical Analysis Plan

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

|---|---|---|---|
| JSS-DM-BIS-01 | Current version Number 1.0 | r revious version number. None | Document Date:00NO v 2019 |

Table 14.3.1.7 Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) by Resolution-Safety Population (N=)

| System Organ Class | Preferred Term | Outcome | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | | |
| SOC 1 | ANY | | | | |
| | PT1 | | | | |
| | | Resolved | | | |
| | | Resolved with Sequelae | | | |
| | | Chronic Condition | | | |
| | | Unknown | | | |
| | | Fatal | | | |
| | PT2 | | | | |
| | 1 12 | Resolved | | | |
| | | Resolved with Sequelae | | | |
| | | Chronic Condition | | | |
| | | Unknown | | | |
| | | Fatal | | | |
| | ••••• | | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator.

**General Note:** 

Protocol No. CPI-CL-022

Confidential

06Nov2019

# Cumberland Pharmaceuticals Inc. JSS Medical Research India Private Limited Data Management Title: Statistical Analysis Plan SOP Number: JSS-DM-BIS-01 Current Version Number1.0 Previous Version Number:None Document Date:06NOV2019

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events] will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

| Cumberland<br>Pharmaceuticals Inc. | | earch India Private Limited<br>a Management | RESPONSIVE RELIABLE RESULTS |
|---|---|---|---|
| Title: S | Title: Statis | stical Analysis Plan | |
| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

#### 14.3.2 SERIOUS ADVERSE EVENTS

Table 14.3.2.1 Summary of Overall Serious Adverse Events -Safety Population (N=)

| | | | D (1 4 (N) ) (1 (D (1) |
|---|---|---|---|
| Category | Parameter, n (%) [1] | Events (N=) | Patients (N=) % of Patien |
| TOTAL<br>Event Occurred | | | |
| | Hospital | | |
| | Home | | |
| | Rehabilitation Facility | | |
| | Outpatient Diagnostic Facility | | |
| | Ambulatory Surgical Facility | | |
| | Outpatient Treatment Facility | | |
| | Other | | |
| Outcome | | | |
| | Death | | |
| | Life-threatening | | |
| | Hospitalization - Initial or Prolonged | | |
| | Other Serious (important Medical Condition) | | |
| | Disability or Permanent Damage | | |
| | Congenital Anomaly/Birth Defect | | |
| subject discontinued | | | |
| Protocol No. CPI-CL-022 | 2 | Confidential | 06Nov2019 |

Statistical Analysis Plan

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

| SOP Number: | | | |
|---|---|---|---|
| JSS-DM-BIS-01 | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |

| Category | Parameter, n (%) [1] | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|
| | Yes | | | |
| | No | | | |
| | Not Applicable | | | |
| Event Abated after the IMP was stopped? | | | | |
| | Yes | | | |
| | No | | | |
| | Not Applicable | | | |
| Event reappeared after IMP reintroduction? | | | | |
| | Yes | | | |
| | No | | | |
| | Not Applicable | | | |
| Was the event expected? | | | | |
| | Expected | | | |
| | Unexpected | | | |

Source Data: Listing 16.2.7.1

Note

[1] Percentages will be calculated using respective column header counts as denominator.

#### **General Note**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events] will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0 (0.0%) [0]".

Protocol No. CPI-CL-022 Statistical Analysis Plan

Confidential

06Nov2019

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

|---|---|---|---|
| JSS-DM-BIS-01 | Current version Number 1.0 | 1 Tevious version number. None | Document Date.00110 V 2019 |

Table 14.3.2.2. Summary of Serious Adverse Events by System Organ Class (SOC) and Preferred Term (PT) -Safety Population (N=)

| System Organ Class | Preferred Term, n(%) [1] | Events (N=) | Patients (N=) | % of Patients |
|---|---|---|---|---|
| TOTAL (ALL SOC/PT) | NA | | | |
| SOC 1 | ANY | | | |
| | PT1 | | | |
| | PT2 | | | |
| SOC 2 | ANY | | | |
| | PT1 | | | |
| | PT2 | | | |

Source Data: Listing 16.2.7.1

Note:

[1] Percentages will be calculated using respective column header counts as denominator.

NA: Not Applicable.

#### **General Note:**

- Adverse events will be coded using MedDRA version 21.1 or later.
- For each SOC and preferred term the number of subjects (percent of subjects) [number of events will be presented.
- Subjects may have reported more than one event per system organ class or preferred term. Subjects will be only counted once for each system organ class or preferred term.
- Zero frequencies will be presented by "0(0.0%) [0]".
- SAE's: Serious Adverse Events

### JSS Medical Research India Private Limited Data Management



#### Title: Statistical Analysis Plan

SOP Number:
JSS-DM-BIS-01

Current Version Number1.0


Document Date:06NOV2019

#### 14.3.3 CONCOMITANT MEDICATION

Table 14.3.3.1 Summary of Concomitant Medication -Safety Population (N=)

| Therapeutic Class | Generic name, n (%) [1] | Overall(N=) |
|---------------------|-------------------------|-------------|
| Therapeutic Class 1 | Any | |
| | Generic Name 1 | |
| | Generic Name 2 | |
| Therapeutic Class 1 | Any | |
| | Generic Name 1 | |
| | Generic Name 2 | |

Source Data: Listing 16.4.4

Note:

#### General Note:

• NA: Not Applicable

<sup>[1]</sup> Percentages will be calculated by taking respective column header group count as denominator.

<sup>•</sup> All Concomitant medications were coded and summarized according to their generic drug names using the WHO Drug classifications version 1st September 2018 or later. One patient may have taken more than one medication.

#### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number: | Compart Warrian North and O | Dunning Verging Namehan Name | Decomposed DetectONOV2010 |
|---|---|---|---|
| JSS-DM-BIS-01 | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |

#### 1.2 LISTINGS

#### 16.2 PATIENT DATA LISTINGS

**Listing 16.2.1 Listing of Patient Study Completion Status** 

| Site No./ Subject No. Age/Gender | | Subject Completed the<br>Study | If Yes, date of study<br>completion/pre-mature<br>discontinuation | Primary reason for<br>pre-mature<br>discontinuation | Other Specify |
|---|---|---|---|---|---|
| XX/NNN | NN/XX | Yes/No | DDMMMYYYY | XX | XX |
| XX/NNN | NN/XX | Yes/No | DDMMMYYYY | XX | XX |
| XX/NNN | NN/XX | Yes/No | DDMMMYYYY | XX | XX |
| | ••• | ••• | ••• | ••• | ••• |

| Did the subject<br>experience any<br>adverse events<br>during the post-<br>treatment period? | Subject's Clinical<br>outcome at the time<br>of the final follow-<br>up | If deceased, date of<br>death | If deceased, cause of<br>death | Did the subject<br>receive NSAIDs or<br>acetaminophen<br>from 4 hours prior<br>to IMP through<br>Study Hour 48? | If Yes, date of<br>restricted<br>Medication | If Yes, Time of<br>restricted<br>Medication |
|---|---|---|---|---|---|---|
| Yes/No | NN/XX | DDMMMYYYY | XX | Yes/No | DDMMMYYYY | XX |
| Yes/No | NN/XX | DDMMMYYYY | XX | Yes/No | DDMMMYYYY | XX |
| Yes/No | NN/XX | DDMMMYYYY | XX | Yes/No | DDMMMYYYY | XX |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

|---|---|---|---|
| JSS-DM-BIS-01 | Current version rumber 1.0 | 1 revious version runnoer.rvone | Document Date:00110 V2017 |

**Listing 16.2.2 Listing of Protocol Deviation** 

| Site No./ | Age/Gender | Visit | Date | Deviation | Comments |
|-------------|------------|-------|-----------|-----------|----------|
| Subject No. | | | | | |
| XX/NNN | NN/XX | XXX | DDMMMYYYY | XX | XX |
| XX/NNN | NN/XX | XXX | DDMMMYYYY | XX | XX |
| XX/NNN | NN/XX | XXX | DDMMMYYYY | XX | XX |
| ••• | ••• | ••• | ••• | ••• | ••• |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

|---|
| JSS-DM-BIS-01 |

**Listing 16.2.3 Listing of Informed Consent** 

| Site ID/ Subject | Age/Gender | Screening Number | Randomization | Date of Screening | Date Informed | Time Informed |
|---|---|---|---|---|---|---|
| No. | | | Number | | Consent Signed | Consent Signed |
| XXX/NNN | NN/XXX | NNN | NNN | DDMMMYYYY | DDMMMYYYY | HH:MM |
| XXX/NNN | NN/XXX | NNN | NNN | DDMMMYYYY | DDMMMYYYY | HH:MM |
| XXX/NNN | NN/XXX | NNN | NNN | DDMMMYYYY | DDMMMYYYY | HH:MM |
| | | ••• | | | | ••• |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

|---|
| JSS-DM-BIS-01 |

Listing 16.2.4 Listing of Inclusion/Exclusion Criteria

| Site ID/Subject No. | Age/Gender | All Inclusion<br>Criteria Met | If No, Inclusion<br>Criteria Number(s) | Exclusion Criteria<br>Met | If Yes, Exclusion Criteria Number(s) | Subject is eligible for the study |
|---|---|---|---|---|---|---|
| XX/NNN | NN/XX | Yes/No | NN | Yes/No | NN | Yes/No |
| XX/NNN | NN/XX | Yes/No | NN | Yes/No | NN | Yes/No |
| XX/NNN | NN/XX | Yes/No | NN | Yes/No | NN | Yes/No |

Statistical Analysis Plan 

#### 

#### **16.2.5 LISTING OF DEMOGRAPHICS**

Listing 16.2.5.1 Listing of Demographics at Screening

| Site ID/Subject No. | Age/Gender | Date of birth | Ethnicity | Race | If race is Multi-<br>racial | Weight (Kg) |
|---|---|---|---|---|---|---|
| XX/NNN | NN/XX | DDMMMYYYY | XX | XX | XX | XX |
| XX/NNN | NN/XX | DDMMMYYYY | XX | XX | XX | XX |
| XX/NNN | NN/XX | DDMMMYYYY | XX | XX | XX | XX |
| ••• | ••• | ••• | •••• | •••• | •••• | •••• |

### JSS Medical Research India Private Limited Data Management



06Nov2019


#### **Title: Statistical Analysis Plan**

|---|---|---|---|
| JSS-DM-BIS-01 | Current version rumber 1.0 | 1 Tevious version ivamoet. Ivone | Bocument Bate.00110 72017 |

**Listing 16.2.5.2 Listing of Medical History** 

| Site<br>ID/Subject | Age/Gender | Condition/<br>Surgery | Generic<br>Name | Therapeutic<br>Class | Onset Date | End Date | Comment | Allergies or reaction |
|---|---|---|---|---|---|---|---|---|
| No.<br>XX/NNN | NN/XX | Yes/No | XX | XX | DDMMMYYYY | DDMMMYYYY | XX | XX |
| XX/NNN | NN/XX | Yes/No | XX | XX | DDMMMYYYY | DDMMMYYYY | XX | XX |
| XX/NNN<br> | NN/XX | Yes/No | XX<br> | XX<br> | DDMMMYYYY | DDMMMYYYY | XX<br> | XX<br> |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number: | | | |
|---|---|---|---|
| | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
| JSS-DM-BIS-01 | | | |

#### 16.2.6 LISTING OF SAFETY ANALYSIS

#### **Listing 16.2.7.1 Listing of Adverse Event**

| Site<br>No./<br>Subjec<br>t No. | Age/Gen<br>der | AE<br>Ter<br>m | Syste<br>m<br>Orga<br>n<br>Class | Preferre<br>d Term | Stop Date | Intens<br>ity | Serio<br>us<br>AE | Resolution:<br>Is the event<br>going? | Resolutio<br>n Date | Resoluti<br>on | IMP<br>Actio<br>n | Event<br>Actio<br>n | Other<br>specif<br>y | Relationship<br>of the event<br>to the IMP |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX/N<br>NN | NN/XX | XX<br>X | XX | XXX | DDMMM<br>YYYY | XX | XX | Yes/No | DDMMM<br>YYYY | XX | XXX | XXX | XXX | XXX |
| XX/N<br>NN | NN/XX | XX<br>X | XX | XXX | DDMMM<br>YYYY | XX | XX | Yes/No | DDMMM<br>YYYY | XX | XXX | XXX | XXX | XXX |
| XX/N<br>NN | NN/XX | XX<br>X | XX | XXX | DDMMM<br>YYYY | XX | XX | Yes/No | DDMMM<br>YYYY | XX | XXX | XXX | XXX | XXX |
| | ••• | | | | ••• | | | | | | | | | |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
|---|---|---|---|
| 199-DM-DI9-01 | | | |

#### 16.2.8 LABORATORY TEST

#### **Listing 16.2.8.1 Listing of Coagulation Assessment**

| Site No./<br>Subject<br>No. | Age/<br>Gender | Visit | If Yes, Date Sample<br>Collected | Time Sample Collected | Lab Test | Result | Result is<br>CS/NCS |
|---|---|---|---|---|---|---|---|
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| | | | ••• | ••• | | | |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |
|---|---|---|---|

Listing 16.2.8.2 Listing of Haematology

| Site No./<br>Subject<br>No. | Age/<br>Gender | Visit | If Yes, Date Sample<br>Collected | Time Sample<br>Collected | Lab Test | Result | Result is<br>CS/NCS |
|---|---|---|---|---|---|---|---|
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | нн:мм | XX | XX | XX |
| | | | ••• | | ••• | | |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

|---|---|---|---|
| JSS-DM-BIS-01 | Current version rumber 1.0 | 1 Tevious version ivamoet. Ivone | Bocument Bate.00110 72017 |

**Listing 16.2.8.3 Listing of Chemistry** 

| Site No./<br>Subject<br>No. | Age/<br>Gender | Visit | If Yes, Date Sample<br>Collected | Time Sample<br>Collected | Lab Test | Result | Result is<br>CS/NCS |
|---|---|---|---|---|---|---|---|
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |
| XX/ NNN | NN/ XX | XX | DDMMMYYYY | HH:MM | XX | XX | XX |

| Cumberland<br>Pharmaceuticals Inc. | JSS Medical Reso<br>Data | RESPONSIVE RELIABLE RESULTS | |
|---|---|---|---|
| | Title: Statistical Analysis Plan | | |
| SOP Number:<br>JSS-DM-BIS-01 | Current Version Number1.0 | Previous Version Number:None | Document Date:06NOV2019 |

#### 16.4 INDIVIDUAL PATIENT DATA LISTINGS

Listing 16.4.1 Listing of Treatment Period IMP Dose 1 and Assessments

| Site No./<br>Subject<br>No. | Age/<br>Gender | Dose Date | Dose Time | IMP/ PRN | Location | Dose administered | If No, Specify | Did the subject receive<br>any PRN Dose of the<br>study drug during the<br>Treatment Period? |
|---|---|---|---|---|---|---|---|---|
| XX/ NNN | NN/ XX | DDMMMYYYY | HH:MM | | NN | Yes/No | XXX | NN |
| XX/ NNN | NN/ XX | DDMMMYYYY | HH:MM | | NN | Yes/No | XXX | NN |
| XX/ NNN | NN/ XX | DDMMMYYYY | HH:MM | | NN | Yes/No | XXX | NN |
| | | ••• | ••• | | | ••• | ••• | ••• |

## Cumberland Pharmaceuticals Inc. JSS Medical Research India Private Limited Data Management Title: Statistical Analysis Plan

Current Version Number 1.0

SOP Number:

JSS-DM-BIS-01

Listing 16.4.2 Listing of Physical Examination


Document Date:06NOV2019

| Site No./ | Age/ Gender | Date of Examination | Time of Examination | Body | Normal/Abnormal | Specify, If |
|---|---|---|---|---|---|---|
| Subject No. | | | | System | | abnormal |
| XX/ NNN | NN/ XX | DDMMMYYYY | HH:MM | XXX | Yes/No | XXX |
| XX/ NNN | NN/ XX | DDMMMYYYY | HH:MM | XXX | Yes/No | XXX |
| XX/ NNN | NN/ XX | DDMMMYYYY | HH:MM | XXX | Yes/No | XXX |
| | | ••• | ••• | | ••• | |

Statistical Analysis Plan 

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| CODNI 1 | | | |
|---|---|---|---|
| JSS-DM-BIS-01 | Current version runnber 1.0 | 1 Tevious version Tumber. Trone | Document Date:00110 12017 |

**Listing 16.4.3 Listing of Vital Signs** 

| Site No./ | Age/ | Visit | Date Performed | Time | Temperature | Route of | Heart Rate | Respiratory | <b>Blood Pressure</b> |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Gender | | | Performed | | Temperature | | Rate | (Systolic /Diastolic) |
| No. | | | | | | Measurement | | | |
| XX/ | NN/ XX | XXX | DDMMMYYYY | HH:MM | NN | XXX | NN | NN | NN/NN |
| NNN | | | | | | | | | |
| XX/ | NN/ XX | XXX | DDMMMYYYY | HH:MM | NN | XXX | NN | NN | NN/NN |
| NNN | | | | | | | | | |
| XX/ | NN/ XX | XXX | DDMMMYYYY | HH:MM | NN | XXX | NN | NN | NN/NN |
| NNN | | | | | | | | | |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

| SOP Number: | | | |
|---|---|---|---|
| SOI Italioon. | Current Version Number 1.0 | Previous Version Number:None | Document Date:06NOV2019 |
| ISS-DM-BIS-01 | Current version reamours. | Trevious version reamoer:reame | Bocament Bate:001(0 (201) |

**Listing 16.4.4 Listing of Concomitant Medication** 

| Site | Age/Ge | Name | Gen | Therap | Do | Dos | If | Dose | If | Ro | If | Was | Start | Star | Ong | End Date | End |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No./ | nder | of | eric | eutic | se | e | Oth | Frequ | Oth | ute | Oth | conco | Date | t | oing | | Tim |
| Subj | | Medic | Nam | Class | | (Un | er, | ency | er, | | er, | mitant | | time | | | e |
| ect | | ation | e | | | its) | spe | | spe | | spe | medica | | | | | |
| No. | | | | | | | cify | | cify | | cify | tion | | | | | |
| | | | | | | | | | | | | prescri | | | | | |
| | | | | | | | | | | | | bed to | | | | | |
| | | | | | | | | | | | | treat | | | | | |
| | | | | | | | | | | | | an | | | | | |
| | | | | | | | | | | | | Advers | | | | | |
| | | | | | | | | | | | | e | | | | | |
| | | | | | | | | | | | | Event? | | | | | |
| XX/ | NN/XX | XXX | XX | XXX | N | XX | XX | XXX | XX | XX | XX | Yes/No | DDMMM | HH: | XXX | DDMMM | HH: |
| NNN | | | X | | N | X | X | | X | X | X | | YYYY | MM | | YYYY | MM |
| XX/ | NN/XX | XXX | XX | XXX | N | XX | XX | XXX | XX | XX | XX | Yes/No | DDMMM | HH: | XXX | DDMMM | HH: |
| NNN | | | X | | N | X | X | | X | X | X | | YYYY | MM | | YYYY | MM |
| XX/ | NN/XX | XXX | XX | XXX | N | XX | XX | XXX | XX | XX | XX | Yes/No | DDMMM | HH: | XXX | DDMMM | HH: |
| NNN | | | X | | N | X | X | | X | X | X | | YYYY | MM | | YYYY | MM |
| | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | | | | ••• | | |

### JSS Medical Research India Private Limited Data Management



#### **Title: Statistical Analysis Plan**

|---|---|---|---|
| JSS-DM-BIS-01 | Current Version Number 1.0 | r revious version number. None | Document Date.00110 v 2019 |

Listing 16.4.5 Listing of Pharmacokinetic Sampling

| Site No./<br>Subject No. | Age/Gender | Time of PK<br>Collection | Date of PK<br>Collection | Collected by means | Date and time the sample spun | Date and time the sample frozen | Number of<br>Aliquot<br>Tubes |
|---|---|---|---|---|---|---|---|
| XX/NNN | NN/XX | HH:MM | DDMMMYYYY | XXX | YYYYMMDD/HH:MM | YYYYMMDD/HH:MM | XXX |
| XX/NNN | NN/XX | HH:MM | DDMMMYYYY | XXX | YYYYMMDD/HH:MM | YYYYMMDD/HH:MM | XXX |
| XX/NNN | NN/XX | HH:MM | DDMMMYYYY | XXX | YYYYMMDD/HH:MM | YYYYMMDD/HH:MM | XXX |
| ••• | •••• | •••• | •••• | •••• | •••• | •••• | •••• |